CLINICAL TRIAL: NCT05829538
Title: The Effect of Sujok and Massage on Pain and Quality of Life in Women With Primary Dysmenorrhea: A Single-Blind, Randomized Controlled Study
Brief Title: SuJok Massage Dismenorea Painful Menstruation
Acronym: SuJok Massage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Halic University (Other)
Collaborators: Tülay Yılmaz (Unknown); Hüsniye Dinç Kaya (Unknown); Sevil Günaydın (Unknown); Zülfiyye Nuraliyeva (Unknown)
Responsible Party: Principal Investigator, Fatma Şule Bilgiç, Lecturer, Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SuJok
Record Dates: First submitted 2023-03-31; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Gynecologic Nursing
Keywords: Su Jok; Massage; Primary Dismenorea; Pain
MeSH Terms: conditions — Pain | interventions — Massage

STUDY DESIGN:
Intervention Model Description: Single Blind Randomized Controled Trials
Who Masked: Participant
Masking Description: In the study, the women were blind to each other in terms of practice and the data evaluator was blinded to the groups in the study in terms of analysis and reporting. Su Jok and massage application and follow-up were carried out by the researcher (FŞB), who could not be blinded to the applications. Randomization was done by another researcher (ZN). In order to avoid bias, the investigator (FSB) did not participate in any step of the pre-test, post-test and statistical evaluation process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Su Jok (Experimental): Su Jok Experimental Group (A): In this study, the seed therapy technique was applied using live buckwheat seeds. Hands were used because it was reported in the literature that hands were used for gynecological pain and were more suitable (Şimşek and Alpar, 2022). The acupuncture point, which is the reflection of the painful area, was determined on the women's hands. This point was massaged for a few minutes by the researcher, and then the buckwheat seed was fixed to this point with a bandage and the area where the seed was applied was massaged for 30 minutes. After each application, VAS evaluation was taken from the women. Su Jok was applied to women in the first three days of menstruation for three cycles.
  Interventions: Behavioral: SuJok
- Massage (Experimental): Experimental Group (B) classical massage techniques (eufluorage, petrissage, friction, tapotman, vibration) was used. Massage was attempted for a total of 20 minutes, 10 minutes on the back and waist, and 10 minutes on the abdominal region, in the first three days of the three cycles. Massage application was started from the back and waist region. Efflorage, petrissage, friction, vibration, taputman and efflorage for one minute were applied to this area, respectively. Afterwards, three minutes of efflorage, petrissage, friction, and one-minute efflorage were applied to the abdominal region, respectively. Odorless, lubricating gel was used during the application. After each application, VAS evaluation was taken from the women. The women were massaged in the first three days of menstruation for three cycles.
  Interventions: Behavioral: Massage
- Control (No Intervention): VAS evaluation was taken on the first three days during three cycles.

INTERVENTIONS:
Behavioral: SuJok — Data were obtained by applying the Su Jok Efficiency Visual Analog Scale (VAS), Functional and Emotional Dysmenorrhea (Painful Menstruation) Scale, and SF-36 Quality of Life Scale.
  Arms: Su Jok
Behavioral: Massage — Data were obtained by applying the Su Jok Efficiency Visual Analog Scale (VAS), Functional and Emotional Dysmenorrhea (Painful Menstruation) Scale, and SF-36 Quality of Life Scale
  Arms: Massage

SUMMARY:
A single-blind randomized controlled study was conducted with female students studying at a foundation university. Women who met the sample selection criteria were randomized into three groups, 40 women in each group, a total of 120 women: Su Jok (A), Massage (B), and Control Group (C). Data were obtained by applying the Data Collection Form, the Visual Analogue Scale (VAS), the Functional and Emotional Dysmenorrhea (Painful Menstruation) Scale, and the SF-36 Quality of Life Scale to the women followed for three menstrual cycles.

DETAILED DESCRIPTION:
This study was performed in a single-blind, randomized controlled type to examine the effect of Su Jok and massage on pain and quality of life in women with primary dysmenorrhea.The sample size in this study was G*Power 3.1.9.2. In the program, 5% first type error, 0.30 standardized effect size, 1:1 distribution ratio, 80% power, and the minimum sample size required for the three groups were calculated as 111 women and 37 women for each group. Considering that there may be losses, 40 women and a total of 120 women were randomized to each group.

"Data Collection Form", "Visiual Analog Scale (VAS)", "Functional and Emotional Dysmenorrhea (Painful Menstruation) Scale", "SF-36, Quality of Life Scale" were used to obtain data.Intervention and Data Collection Stage 1: VAS was applied to the women who volunteered to participate in the study on the first day of menstruation, and women with a mean score of 5 and above and meeting the sample selection criteria were randomized into three separate groups as A, B, and C. The researcher who performed the randomization ensured that the women were assigned to the control and experimental groups and did not share this information with the other researchers. Data Collection Form, Functional and Emotional Dysmenorrhea (Painful Menstruation) Scale, SF-36 Quality of Life Scale were applied to all women on the first day of the next menstruation. Since the data collection tools were based on self-report, the woman was allowed to answer in a calm environment and alone. The environment where the applications will be held was arranged in such a way that the researcher and the participant could sit opposite each other with two chairs and an application table. Entry and exit to the room was prevented until the application was over. The environment was quiet.

Stage 2 Su Jok Experimental Group (A): In this study, the seed therapy technique was applied using live buckwheat seeds. Hands were used because it was reported in the literature that hands were used for gynecological pain and were more suitable.The acupuncture point, which is the reflection of the painful area, was determined on the women's hands. This point was massaged for a few minutes by the researcher, and then the buckwheat seed was fixed to this point with a bandage and the area where the seed was applied was massaged for 30 minutes. After each application, VAS evaluation was taken from the women. Su Jok was applied to women in the first three days of menstruation for three cycles.Experimental Group (B) to whom massage was applied: Massage application determined by scanning the literature and taking expert opinion classical massage techniques (eufluorage, petrissage, friction, tapotman, vibration) was used. Massage was attempted for a total of 20 minutes, 10 minutes on the back and waist, and 10 minutes on the abdominal region, in the first three days of the three cycles. Massage application was started from the back and waist region. Efflorage, petrissage, friction, vibration, taputman and efflorage for one minute were applied to this area, respectively. Afterwards, three minutes of efflorage, petrissage, friction, and one-minute efflorage were applied to the abdominal region, respectively. Odorless, lubricating gel was used during the application. After each application, VAS evaluation was taken from the women. Massage was applied to the women in the first three days of menstruation for three cycles.

Control Group (C): VAS assessment was obtained for the first three days during three cycles.

Stage 3 Functional and Emotional Dysmenorrhea (Painful Menstruation) Scale and SF-36 Quality of Life Scale were applied to all women included in the study on the third day of the third cycle.

ELIGIBILITY:
Inclusion Criteria:

* Not diagnosed with chronic and mental illness,
* Not using hormonal contraceptives and analgesics,
* Not having a pregnancy history, d) having regular menstrual cycles in the last 6 months (bleeding between 3-8 days and 21-35 days)
* Verbal Women who stated that they had dysmenorrhea
* 18-35 years old g) Women who defined menstrual pain as 5 or higher according to the Visual Analogue Scale (VAS) were included.

Exclusion Criteria:

* Dysmenorrhea and a gynecological diagnosis,
* Regular exercise, massage and Su Jok practices were not included.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with painful menstruation
Enrollment: 120 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Menstrual Pain VAS | 12 Weeks
  The effect of the intervention on menstrual pain was measured by VAS
Affected by dysmenorrhea | 12 Weeks
  Measured with the Functional and Emotional Dysmenorrhea (Painful Menstruation) Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data Collection: 4 Months Analysis: 3 Months Reporting and Publication 4 Months